CLINICAL TRIAL: NCT02348970
Title: Multicenters, Randomised Clinical Trial, to Evaluate Efficacy and Compliance of Mandibular Advancement Devices ONIRIS® vs. Laboratory Devices TALI in Patients With Syndrome of Obstructive Sleep Apnea and Hypopneas
Brief Title: Efficacy and Compliance of the Mandibular Advancement Devices ONIRIS® vs. Custom Made Devices
Acronym: IRIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ONIRIS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONI-003
Record Dates: First submitted 2015-01-12; First posted 2015-01-28 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: mandibular advancement devices ONIRIS®; obstructive sleep apnea and hypopneas
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mandibular advancement devices ONIRIS® (Experimental): The patients will use the mandibular advancement devices ONIRIS®
  Interventions: Device: ONIRIS®
- laboratory devices TALI (Active Comparator): The patients will use the laboratory devices TALI
  Interventions: Device: TALI

INTERVENTIONS:
Device: ONIRIS® — sleeping test
  Arms: mandibular advancement devices ONIRIS®
Device: TALI — sleeping test
  Arms: laboratory devices TALI

SUMMARY:
To evaluate the efficacy (non-inferiority) in terms of response between patients using custom fitted mandibular advancement devices ONIRIS® and patient using laboratory custom made devices TALI, after 2 months of use. Sleeping tests were performed.

DETAILED DESCRIPTION:
Open, non-inferiority, controlled and rndomised clinical trial. Six months of inclusion. Each included patient will be followed during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe syndrome of obstructive sleep apnea and hypopneas refusing or withdrawal from continuous positive pression ventilation
* no dental, paro-dental or articular contraindication
* patients never treated by mandibular advancement devices

Exclusion Criteria:

* severe psychiatric or neuromuscular disorders appreciated by the investigator
* more than 20% of apneas and central hypoapneas
* severe syndrome of obstructive sleep apnea and hypopneas with IAH > 30% associated with another sleeping pathology
* BMI > 30kg/m2
* patient with an uncontrollable nausea reflex
* epileptic patients
* pregnant patients
* patient without written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacity (non-inferiority) in terms of response between patients using mandibular advancement devices ONIRIS® and patient using devices produced in a laboratoryTALI after 2 months of use. | 2 monthes of use
  The response to the treatment is defined as:
  * complete patient response: AHI per hour of sleep < 10 or
  * partial patient response: AHI per hour of sleep reduced by 50% at visit M2 compared to baseline

SECONDARY OUTCOMES:
Evolution of AHI, AI and HI | at M2 and at M12
  AHI per hour of sleep with the same modalities as the one used for diagnosis (realised by ambulatory PG or PSG)
Percentage of patients responder | at M2 and M12
  Percentage of patients responder at the last control exam
Evolution during the study of the principal criteria concerning the sleep | at baseline, M2, M6 and M12
  Snoring measured by VAS, Epworth Sleepness Scale measuring daytime sleepness, Pichot Questionnaire measuring fatigue and depression
Evolution of the quality of life | at baseline, M2, M6 and M12
  Quality of life evaluated by SF12 at each visit
Evolution of the compliance | at M2, M6 and M12
  Percantage of compliance (excellent > 85%, good > 50%)
Evolution of tolerance | at M2, M6 and M12
  Nature, frequency and intensity of AE at each visit
AE and SAE occuring during the study | at M2, M6 and M12
  Description and comparison at each group of AE and SAE
Evolution of arterial hypertension | at baseline, M2, M6 and M12
  Arterial hypertension evaluated at each visit

CONTACTS AND LOCATIONS:
Overall Officials: RAYMOND Nathalie, MD, Principal Investigator — Hôpital Bel Air
Locations (10):
- France (10):
  - Clinique Bel-Air, Bordeaux
  - Polyclinique Saint Privat, Boujan-sur-Libron
  - CHU de Grenoble, La Tronche
  - Hôpital André Mignot, Le Chesnay
  - Medical Practice, Les Pavillons-sous-Bois
  - Medical Practice, Maisons-Alfort
  - CHU Montpellier, Montpellier
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Medical Practice, Perpignan
  - Centre Cardiologique du Nord, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pepin JL, Raymond N, Lacaze O, Aisenberg N, Forcioli J, Bonte E, Bourdin A, Launois S, Tamisier R, Molinari N. Heat-moulded versus custom-made mandibular advancement devices for obstructive sleep apnoea: a randomised non-inferiority trial. Thorax. 2019 Jul;74(7):667-674. doi: 10.1136/thoraxjnl-2018-212726. Epub 2019 May 3. PMID 31053619